CLINICAL TRIAL: NCT01555775
Title: Compared Effect of a Fruit Milk Shake With a Protein-Carbohydrate Supplement on Muscle Damage, Inflammation, Oxidative Stress and Functional Recovery, After Resistance Exercise
Brief Title: Compared Effect of a Fruit Milk Shake With a Protein-Carbohydrate Supplement on Recovery After Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Monica Sousa, Principal Investigator, BSc, Universidade do Porto
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: SFRH/BD/75276/2010
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Muscle Damage; Inflammation; Oxidative Stress; Functional Recovery
Keywords: exercise-induced muscle damage; nutritional recovery; nutritional supplement; natural food
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- P-CHO supplement (Experimental): This group will drink the P-CHO supplement in the first trial and the fruit milk shake in the second.
  Interventions: Dietary Supplement: P-CHO supplement
- Fruit Milk Sake (Experimental): This group will drink the fruit milk shake in the first trial and the P-CHO supplement in the second.
  Interventions: Dietary Supplement: Fruit Milk Shake

INTERVENTIONS:
Dietary Supplement: P-CHO supplement — In the first trial, this group will drink a protein (P)-carbohydrate (CHO) supplement and in the second trial the fruit milk shake.
  Other Names: Available in a common local market.
  Arms: P-CHO supplement
Dietary Supplement: Fruit Milk Shake — The fruit content of the milk shake will be 100 g of strawberry and the amount of banana necessary to guaranty 0.8-1.2 g CHO • kg-1 BW • h-1.
  Other Names: Strawberry, bananas, skimmed milk
  Arms: Fruit Milk Sake

SUMMARY:
The aim of this study is to assess the effect of ingesting a commercial carbohydrate and protein dietary supplement in powder form (P-CHO supplement) or a milk shake with skimmed milk, strawberries and banana (MS), after resistance exercise, in muscle damage, oxidative stress, inflammation and functional recovery. It is hypothesised if the ingestion of a milk shake with skimmed milk and fruit (strawberry and banana) has the same impact on markers of muscle damage, oxidative stress, inflammation and functional recovery induced by resistance exercise, as the intake of a commercial powder with the same CHO and protein amounts.

Fifteen adult athletes from the Portuguese Athletic Federation will complete 2 trials separated at least by 2 weeks. Alternate legs and drinks will be used in each trial and participants will be overnight-fasted. This study will have a single-blind, randomized, crossover, repeated-measures experimental design. In each trial, after warm-up, the eccentric peak torque of the knee joint extensors will be determined using an isokinetic dynamometer. After this, participants will complete an isokinetic exercise until exhaustion at a constant angular velocity of 60° • s-1. After the exhaustion protocol, athletes will perform again the peak torque determination. Immediately after, participants will drink the P-CHO supplement or MS during the first 2 h. Both drinks will contain 0.8-1.2 g carbohydrates • kg-1 • h-1 and 0.2-0.4 g protein • kg-1 • h-1. Twenty four and 48 h after the exhaustion protocol participants will return to the laboratory to repeat the peak torque determination. Blood samples will be collected before warming-up, immediately and 2 h after the last peak torque determination and 24 h and 48 h after. Serum samples will be analyzed for creatine kinase, lactate dehydrogenase, interleukine-6, protein carbonyls and total antioxidant status. The delayed onset muscle soreness, using a visual analogue scale, and girths will be measured at the same moments as blood sampling. Two-way repeated-measures ANOVA will be used for statistical analysis of the data.

DETAILED DESCRIPTION:
Sample:

Fifteen adult athletes from the Portuguese Athletic Federation will be invited to participate in this study. They must be healthy and lactose tolerant. Athletes will be voluntary and should receive an explanatory document with the aims of the study. They must also sign an informed consent to participate. To help ensuring that the metabolic conditions are similar between trials, subjects will be instructed to fulfill a food record and a physical activity record of the 2 days prior to each trial (Shirreffs, Watson, & Maughan, 2007). It will be asked not to make drastic changes in diet and to avoid strenuous exercise during this period.

Experimental Protocol:

This study will have a single-blind, randomized, crossover, repeated-measures experimental design. As shown in Figure 1, each participant should complete 2 trials, with a wash out period of, at least, 2 weeks. In one trial subjects will randomly drink the P-CHO supplement and in the other, the MS. In order to minimize any repeated bout effect, different legs will be used in each trial (Howatson et al., 2010).

About one week before the exercise protocol, participants will be familiarized with the experimental procedures and measurements. At this time, anthropometric assessments (BW, height and body fat percentage) will also be taken.

All tests should be performed in the morning, in a fasted state. At the beginning of each trial, the participants will warm-up for 5 min using a cycle ergometer at an intensity of 70-100 rpm. After the warm-up, the eccentric peak torque of the knee joint extensors muscles will be determined by isokinetic dynamometry (Biodex®, system IV). Then, the participants will complete concentric/eccentric knee extension/flexion exercise protocol until exhaustion. After exhaustion, eccentric peak torque determination will be repeated. Immediately after finishing the isokinetic test, participants will drink the P-CHO supplement or MS during the first 2 hours post-exercise. The drinks will be taken in 2 bolus per hour, during 2 h. During the 2 days after the exhaustion protocol (24 h and 48 h after), participants will return to the laboratory to repeat eccentric peak torque determination after a similar warm-up of the day before.

Drinks' Composition:

The nutritional formula of both drinks will be equal in terms of CHO and protein content in order to achieve the recommendation values of 0.8-1.2 g CHO • kg-1 BW • h-1 and 0.2-0.4 g protein • kg-1 BW • h-1 (Beelen et al 2010). They will also have similar amounts of vitamin C.

The fruit content of the MS will be 100 g of strawberry and the amount of banana necessary to guaranty 0.8-1.2 g CHO • kg-1 BW • h-1. Regarding the P-CHO supplement, it has to be available in a common local market and meet the recommend amounts of CHO and protein for the recovery period. If necessary, vitamin C will be added to match the MS content.

Exhaustion Protocol:

For inducting exhaustion, a concentric/eccentric knee extension/flexion exercise until exhaustion will be used. At the first day of each trial, the exhaustion protocol will be conducted. Securely fastened into the test chair of the isokinetic dynamometer with the knee joint of the test limb aligned with the axis of rotation of the dynamometer and the distal lower limb secured to the dynamometer's test arm, subjects will initially complete 3 maximal repetitions of knee joint extension and flexion at a constant angular velocity of 60°•s-1 to determine the subject's maximal peak torque of the knee extensors muscles (the best of the 3 repetitions). After this, the exhaustion protocol it will be conducted. The protocol will consist of 3 bouts of a concentric/eccentric knee extension/flexion exercise, at 60°•s-1, with a 200-second rest time between sets. The first and second set will be composed by 100 repetitions; in the third set, subjects will perform n repetitions until the eccentric peak value of 3 consecutive repetitions fell below 25% of the initial knee extensor eccentric peak torque value. The range of motion will be from 50° to 110° flexion in the knee (0º = full knee extension).

Participants will receive verbal encouragement to perform maximally throughout the exercise protocol.

Functional Recovery:

To monitor force recovery, measures of eccentric peak torque of the knee joint extensor muscles will be determined. Athletes will perform the isokinetic strength tests immediately before and after the exhaustion protocol and 24 and 48 h after the exhaustion protocol, for each trial. The exercise will consist of 3 maximal repetitions to determine eccentric knee joint extension peak torque at a constant angular velocity of 60°•s-1. The range of motion will be similar to the one used in the exhaustion protocol.

Blood Sampling and Biomarkers:

For each trial, blood will be taken from an antecubital vein after the participant arrives at the laboratory, in a fasted state. Blood samples will also be collected immediately after the last peak torque determination and 2, 24 and 48 h after.

The following blood markers will be used:

* Muscle damage: CK and LDH;
* Inflammation: IL-6;
* Oxidative stress: protein carbonyls and TAS.

Other Measurements:

The DOMS and circumferential measurements will be measured at the same moments as blood sampling.

A visual analogue scale (VAS), 10 cm in length, will be used to determine DOMS (Bijur, Silver, & Gallagher, 2001).

The mid-thigh girth measurement will be done according to the anthropometric technique suggested by the International Society for the Advancement of Kinanthropometry (ISAK). Three other girths will be measured: 5, 15 and 25 cm above the superior border of the patella. These measurements will allow monitoring the oedema caused by inflammation.

Body Composition:

Weight and height will be measured according to the methodology proposed by the International Society for the ISAK. It will be calculated the body mass index (BMI) and the percentage of body fat by measuring four skinfolds (biceps, triceps, subscapular and suprailiac) according to the technique proposed by ISAK. The value of the measurements will be converted to body density and using the formula: Durnin and Womersley 1974 (Costa, 2001). Later, the body density value will be converted to percentage of body mass, using the formula of Siri (Costa, 2001).

Dietary Intake:

Athletes will be asked to carry out food records 2 days prior to each trial. Each individual will be informed both orally and in writing, by an expert nutritionist, on their correct completion. It also will be required to register the time and place where food consumption was made. Subsequently, data will be processed through a computer program (Food Processor®) to convert the information into energy and nutrients and calculate mean intakes.

Physical Activity:

Two days prior to each trial, athletes will record the type, intensity and duration of physical activities in registration documents distributed previously.

Statistical Analysis:

Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS 18 for Windows TM®). The results will be expressed as mean ± standard deviation and it will be considered a statistically significant for p < 0.05. Normality will be assessed by the Kolmogorov-Smirnov test. Data will be analyzed by two-way repeated-measures ANOVA (treatment [two levels: MS and P-CHO supplement] vs time [five levels]) to determine whether there are any statistically significant effects of time or treatment (Bowtell, Sumners, Dyer, Fox, & Mileva, 2011). The Mauchly sphericity test will be used to check homogeneity of covariance for all ANOVA analyses; violations of the assumption of sphericity will be correct using the Greenhouse-Geisser adjustment. Where appropriate, the effect size (ƞ2) will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* healthy and lactose tolerant

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Maximal peak torque of the knee extensors muscles | Up to 48 h
  To monitor functional recovery
Creatine kinase | Up to 48 h
  To monitor muscle damage
Lactate dehydrogenase | Up to 48 h
  To monitor muscle damage
Interleukine-6 | Up to 48 h
  To monitor the inflammatory process
Total antioxidant status | Up to 48 h
  To monitor oxidative stress
Delayed onset muscle soreness | Up to 48 h
  By a visual analogue scale, 10 cm in length. To monitor muscle soreness
Mid-thigh girth, Three other girths will be measured: 5, 15 and 25 cm above the superior border of the patella. | Up to 48 h
  To monitor the inflammatory process
Protein carbonyls | Up to 48 h
  To monitor oxidative stress

SECONDARY OUTCOMES:
Percentage of body fat | 1 week before the first trial
Food records | 2 days before each trial
  To assess energy intake (kcal)
Physical activity records | 2 days before each trial
  To assess energy expenditure (kcal)

CONTACTS AND LOCATIONS:
Overall Officials: José Soares, PhD, Study Director — Faculdade de Desporto, Universidade do Porto; Monica V. Sousa, BSc, Principal Investigator — Faculdade de Desporto, Universidade do Porto; Vitor H Teixeira, PhD, Study Chair — Faculdade de Ciências da Nutrição e Alimentação, Universidade do Porto
Locations (1):
- Faculdade de Desporto, Universidade do Porto, Porto, Portugal

REFERENCES:
- [Background] Banerjee AK, Mandal A, Chanda D, Chakraborti S. Oxidant, antioxidant and physical exercise. Mol Cell Biochem. 2003 Nov;253(1-2):307-12. doi: 10.1023/a:1026032404105. PMID 14619981
- [Background] Battino M, Mezzetti B. Update on fruit antioxidant capacity: a key tool for Mediterranean diet. Public Health Nutr. 2006 Dec;9(8A):1099-103. doi: 10.1017/S1368980007668554. PMID 17378947
- [Background] Beelen M, Burke LM, Gibala MJ, van Loon L JC. Nutritional strategies to promote postexercise recovery. Int J Sport Nutr Exerc Metab. 2010 Dec;20(6):515-32. doi: 10.1123/ijsnem.20.6.515. PMID 21116024
- [Background] Ben-Amotz A, Levy Y. Bioavailability of a natural isomer mixture compared with synthetic all-trans beta-carotene in human serum. Am J Clin Nutr. 1996 May;63(5):729-34. doi: 10.1093/ajcn/63.5.729. PMID 8615356
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Bos C, Metges CC, Gaudichon C, Petzke KJ, Pueyo ME, Morens C, Everwand J, Benamouzig R, Tome D. Postprandial kinetics of dietary amino acids are the main determinant of their metabolism after soy or milk protein ingestion in humans. J Nutr. 2003 May;133(5):1308-15. doi: 10.1093/jn/133.5.1308. PMID 12730415
- [Background] Bowtell JL, Sumners DP, Dyer A, Fox P, Mileva KN. Montmorency cherry juice reduces muscle damage caused by intensive strength exercise. Med Sci Sports Exerc. 2011 Aug;43(8):1544-51. doi: 10.1249/MSS.0b013e31820e5adc. PMID 21233776
- [Background] Brancaccio P, Lippi G, Maffulli N. Biochemical markers of muscular damage. Clin Chem Lab Med. 2010 Jun;48(6):757-67. doi: 10.1515/CCLM.2010.179. PMID 20518645
- [Background] Burke LM, Castell LM, Stear SJ. BJSM reviews: A-Z of supplements: dietary supplements, sports nutrition foods and ergogenic aids for health and performance Part 1. Br J Sports Med. 2009 Oct;43(10):728-9. doi: 10.1136/bjsm.2009.063941. No abstract available. PMID 19808984
- [Background] Burke LM, Castell LM, Stear SJ, Rogers PJ, Blomstrand E, Gurr S, Mitchell N, Stephens FB, Greenhaff PL. BJSM reviews: A-Z of nutritional supplements: dietary supplements, sports nutrition foods and ergogenic aids for health and performance Part 4. Br J Sports Med. 2009 Dec;43(14):1088-90. doi: 10.1136/bjsm.2009.068643. No abstract available. PMID 19955167
- [Background] Cao G, Prior RL. Comparison of different analytical methods for assessing total antioxidant capacity of human serum. Clin Chem. 1998 Jun;44(6 Pt 1):1309-15. PMID 9625058
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Close GL, Ashton T, McArdle A, Maclaren DP. The emerging role of free radicals in delayed onset muscle soreness and contraction-induced muscle injury. Comp Biochem Physiol A Mol Integr Physiol. 2005 Nov;142(3):257-66. doi: 10.1016/j.cbpa.2005.08.005. Epub 2005 Sep 8. PMID 16153865
- [Background] Ebbeling CB, Clarkson PM. Exercise-induced muscle damage and adaptation. Sports Med. 1989 Apr;7(4):207-34. doi: 10.2165/00007256-198907040-00001. PMID 2657962
- [Background] Ehlenfeldt MK, Prior RL. Oxygen radical absorbance capacity (ORAC) and phenolic and anthocyanin concentrations in fruit and leaf tissues of highbush blueberry. J Agric Food Chem. 2001 May;49(5):2222-7. doi: 10.1021/jf0013656. PMID 11368580
- [Background] Eston RG, Mickleborough J, Baltzopoulos V. Eccentric activation and muscle damage: biomechanical and physiological considerations during downhill running. Br J Sports Med. 1995 Jun;29(2):89-94. doi: 10.1136/bjsm.29.2.89. PMID 7551767
- [Background] Evans WJ. Vitamin E, vitamin C, and exercise. Am J Clin Nutr. 2000 Aug;72(2 Suppl):647S-52S. doi: 10.1093/ajcn/72.2.647S. PMID 10919971
- [Background] Finaud J, Lac G, Filaire E. Oxidative stress : relationship with exercise and training. Sports Med. 2006;36(4):327-58. doi: 10.2165/00007256-200636040-00004. PMID 16573358
- [Background] Halliwell B. The antioxidant paradox. Lancet. 2000 Apr 1;355(9210):1179-80. doi: 10.1016/S0140-6736(00)02075-4. No abstract available. PMID 10791396
- [Background] Heim KE, Tagliaferro AR, Bobilya DJ. Flavonoid antioxidants: chemistry, metabolism and structure-activity relationships. J Nutr Biochem. 2002 Oct;13(10):572-584. doi: 10.1016/s0955-2863(02)00208-5. PMID 12550068
- [Background] Howatson G, McHugh MP, Hill JA, Brouner J, Jewell AP, van Someren KA, Shave RE, Howatson SA. Influence of tart cherry juice on indices of recovery following marathon running. Scand J Med Sci Sports. 2010 Dec;20(6):843-52. doi: 10.1111/j.1600-0838.2009.01005.x. PMID 19883392
- [Background] Howatson G, van Someren KA. The prevention and treatment of exercise-induced muscle damage. Sports Med. 2008;38(6):483-503. doi: 10.2165/00007256-200838060-00004. PMID 18489195
- [Background] Ivy JL, Goforth HW Jr, Damon BM, McCauley TR, Parsons EC, Price TB. Early postexercise muscle glycogen recovery is enhanced with a carbohydrate-protein supplement. J Appl Physiol (1985). 2002 Oct;93(4):1337-44. doi: 10.1152/japplphysiol.00394.2002. PMID 12235033
- [Background] Jackman SR, Witard OC, Jeukendrup AE, Tipton KD. Branched-chain amino acid ingestion can ameliorate soreness from eccentric exercise. Med Sci Sports Exerc. 2010 May;42(5):962-70. doi: 10.1249/MSS.0b013e3181c1b798. PMID 19997002
- [Background] Jeukendrup AE. Carbohydrate intake during exercise and performance. Nutrition. 2004 Jul-Aug;20(7-8):669-77. doi: 10.1016/j.nut.2004.04.017. PMID 15212750
- [Background] Jeukendrup AE. Carbohydrate and exercise performance: the role of multiple transportable carbohydrates. Curr Opin Clin Nutr Metab Care. 2010 Jul;13(4):452-7. doi: 10.1097/MCO.0b013e328339de9f. PMID 20574242
- [Background] Karlsson HK, Nilsson PA, Nilsson J, Chibalin AV, Zierath JR, Blomstrand E. Branched-chain amino acids increase p70S6k phosphorylation in human skeletal muscle after resistance exercise. Am J Physiol Endocrinol Metab. 2004 Jul;287(1):E1-7. doi: 10.1152/ajpendo.00430.2003. Epub 2004 Mar 2. PMID 14998784
- [Background] Kerksick C, Harvey T, Stout J, Campbell B, Wilborn C, Kreider R, Kalman D, Ziegenfuss T, Lopez H, Landis J, Ivy JL, Antonio J. International Society of Sports Nutrition position stand: nutrient timing. J Int Soc Sports Nutr. 2008 Oct 3;5:17. doi: 10.1186/1550-2783-5-17. PMID 18834505
- [Background] Lamprecht M, Greilberger J, Oettl K. Analytical aspects of oxidatively modified substances in sports and exercises. Nutrition. 2004 Jul-Aug;20(7-8):728-30. doi: 10.1016/j.nut.2004.04.016. PMID 15212757
- [Background] Leeuwenburgh C, Heinecke JW. Oxidative stress and antioxidants in exercise. Curr Med Chem. 2001 Jun;8(7):829-38. doi: 10.2174/0929867013372896. PMID 11375753
- [Background] Maughan RJ, King DS, Lea T. Dietary supplements. J Sports Sci. 2004 Jan;22(1):95-113. doi: 10.1080/0264041031000140581. PMID 14971436
- [Background] McGinley C, Shafat A, Donnelly AE. Does antioxidant vitamin supplementation protect against muscle damage? Sports Med. 2009;39(12):1011-32. doi: 10.2165/11317890-000000000-00000. PMID 19902983
- [Background] Proteggente AR, Pannala AS, Paganga G, Van Buren L, Wagner E, Wiseman S, Van De Put F, Dacombe C, Rice-Evans CA. The antioxidant activity of regularly consumed fruit and vegetables reflects their phenolic and vitamin C composition. Free Radic Res. 2002 Feb;36(2):217-33. doi: 10.1080/10715760290006484. PMID 11999391
- [Background] Roy BD. Milk: the new sports drink? A Review. J Int Soc Sports Nutr. 2008 Oct 2;5:15. doi: 10.1186/1550-2783-5-15. PMID 18831752
- [Background] Sacheck JM, Blumberg JB. Role of vitamin E and oxidative stress in exercise. Nutrition. 2001 Oct;17(10):809-14. doi: 10.1016/s0899-9007(01)00639-6. PMID 11684385
- [Background] Sellappan S, Akoh CC, Krewer G. Phenolic compounds and antioxidant capacity of Georgia-grown blueberries and blackberries. J Agric Food Chem. 2002 Apr 10;50(8):2432-8. doi: 10.1021/jf011097r. PMID 11929309
- [Background] Shirreffs SM, Watson P, Maughan RJ. Milk as an effective post-exercise rehydration drink. Br J Nutr. 2007 Jul;98(1):173-80. doi: 10.1017/S0007114507695543. Epub 2007 Apr 26. PMID 17459189
- [Background] Smith C, Kruger MJ, Smith RM, Myburgh KH. The inflammatory response to skeletal muscle injury: illuminating complexities. Sports Med. 2008;38(11):947-69. doi: 10.2165/00007256-200838110-00005. PMID 18937524
- [Background] Steinberg JG, Delliaux S, Jammes Y. Reliability of different blood indices to explore the oxidative stress in response to maximal cycling and static exercises. Clin Physiol Funct Imaging. 2006 Mar;26(2):106-12. doi: 10.1111/j.1475-097X.2006.00658.x. PMID 16494601
- [Background] Szajdek A, Borowska EJ. Bioactive compounds and health-promoting properties of berry fruits: a review. Plant Foods Hum Nutr. 2008 Dec;63(4):147-56. doi: 10.1007/s11130-008-0097-5. PMID 18931913
- [Background] Urso ML, Clarkson PM. Oxidative stress, exercise, and antioxidant supplementation. Toxicology. 2003 Jul 15;189(1-2):41-54. doi: 10.1016/s0300-483x(03)00151-3. PMID 12821281
- [Background] Verburg E, Murphy RM, Stephenson DG, Lamb GD. Disruption of excitation-contraction coupling and titin by endogenous Ca2+-activated proteases in toad muscle fibres. J Physiol. 2005 May 1;564(Pt 3):775-90. doi: 10.1113/jphysiol.2004.082180. Epub 2005 Mar 3. PMID 15746171
- [Background] Westerblad H, Bruton JD, Allen DG, Lannergren J. Functional significance of Ca2+ in long-lasting fatigue of skeletal muscle. Eur J Appl Physiol. 2000 Oct;83(2-3):166-74. doi: 10.1007/s004210000275. PMID 11104057
- [Background] Yeum KJ, Russell RM, Krinsky NI, Aldini G. Biomarkers of antioxidant capacity in the hydrophilic and lipophilic compartments of human plasma. Arch Biochem Biophys. 2004 Oct 1;430(1):97-103. doi: 10.1016/j.abb.2004.03.006. PMID 15325916
- See also: Web page of the institution that funds the individual Ph.D. grant (SFRH/BD/75276/2010) — http://www.fct.pt/